CLINICAL TRIAL: NCT00994162
Title: A Prospective, Open Labelled, Multicentre Evaluation of the Use of EZCare/V1STA in the Management of Acute and Chronic Wounds
Brief Title: Evaluation of the Use of EZCare/V1STA in the Management of Acute and Chronic Wounds
Acronym: EZCARE/V1STA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIME 012
Record Dates: First submitted 2009-10-09; First posted 2009-10-14 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2020-03

CONDITIONS: Wounds
Keywords: NPWT; Gauze-based filler; Acute or Chronic Wounds; Efficacy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Negative Pressure Wound Therapy (Experimental): Application of NPWT therapy to the wound
  Interventions: Device: EZCare/V1STA Negative Pressure Wound Therapy System

INTERVENTIONS:
Device: EZCare/V1STA Negative Pressure Wound Therapy System — Vacuum Source and dressing kit that generates negative pressure over the wound.
  Other Names: EZCare/V1STA Device and gauze-based filler dressing kit

SUMMARY:
The aim of this evaluation is to assess the performance of the EZCare/V1STA products, in many different clinical environments, in order to gain a greater insight into the effects of this negative pressure wound therapy (NPWT) in a variety of wound types.

DETAILED DESCRIPTION:
Patients meeting the eligibility criteria and agreeing to consent to their participation in the evaluation will receive treatment with the evaluation product for a maximum of 10 dressing changes or up to a maximum of 30 days treatment with the EZCare/V1STA products, whichever comes first. Treatment will commence on Day 0 and dressing changes will take place as deemed appropriate by the Clinician responsible for the patient, however it is recommended that the dressing is changed at least every 3 days in accordance with the product instructions for use.

Treatment will stop when, in the opinion of the Clinician, sufficient wound progress has taken place to merit a change in treatment regime i.e. surgical intervention (e.g. graft) or the use of more traditional dressings. Treatment with the evaluation product will not proceed past 30 days.

Patients will be treated with a pressure setting of between 40mmHg and 80mmHg for the duration of treatment.

A follow up wound assessment will take place 7 days post treatment discontinuation.

If required, debridement may be performed prior to and during the patients participation in this evaluation.

NOTE: While starting out as two individual studies (EZCare CIME 012 and V1STA CIME 010), these studies were ultimately combined and analyzed together as one set of results. The decision to report the two studies with a single Clinical Study Report was due to high levels of similarity in both the study designs and the products themselves; the individual study designs were largely similar with the same patient population criteria, study endpoints, and data capture requirements; and the products were identical in terms of their indications for use and therapeutic delivery of NPWT.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age
* Males and females - provided they are not pregnant and if of reproductive age are using contraception
* The patient must have an acute or chronic wound deemed suitable for treatment with NPWT
* The patient is able to understand the evaluation and is willing to consent to the evaluation

Exclusion Criteria:

* Presence of necrotic tissue or >25% slough in the reference wound. Once debridement has taken place the patient may proceed to enter the evaluation.
* Previously confirmed and untreated osteomyelitis.
* Malignancy in the reference wound bed or margins of the wound.
* Active bleeding in the reference wound. Once haemostasis has been achieved, the patient may proceed to enter the evaluation.
* Exposure of blood vessels or organs at the base of the reference wound.
* Presence of untreated infection in the reference wound. (Infected wounds being treated with systemic antibiotics are permitted)
* Patients with a known history of poor compliance with medical treatment.
* Patients who have participated in this evaluation previously and who healed or were withdrawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond M Dunn, MD, Principal Investigator — UMass Memorial Health
Locations (1):
- UMass Memorial Medical Center, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] Banwell PE, Teot L. Topical negative pressure (TNP): the evolution of a novel wound therapy. J Wound Care. 2003 Jan;12(1):22-8. doi: 10.12968/jowc.2003.12.1.26451. PMID 12572233
- [Background] Luckraz H, Murphy F, Bryant S, Charman SC, Ritchie AJ. Vacuum-assisted closure as a treatment modality for infections after cardiac surgery. J Thorac Cardiovasc Surg. 2003 Feb;125(2):301-5. doi: 10.1067/mtc.2003.74. PMID 12579098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: While starting out as 2 individual studies (EZCare CIME 012 and V1STA CIME 010), these studies were ultimately combined and analyzed together as one set of results. The decision to report the 2 studies with a single CSR was due to high levels of similarity in both the study designs and the products themselves. The study was further divided into subgroups of subjects with a grafted wound site (21 subjects) or subjects with a non-grafted wound site (131 subjects) to compare wound types.
Pre-assignment Details: A total of 153 subjects were enrolled; however, one V1STA subject was withdrawn from the study due to medical complications that prohibited the application of the NPWT system. The subject was excluded from the full analysis set (FAS) population, but included in the safety (SAF) population.
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy
Started | 153
Participants Receiving Treatment | 152
Completed | 125
Not Completed | 28
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2
Not completed — Product Complaint | 1
Not completed — Poor Compliance | 5
Not completed — Lack of Response | 3
Not completed — Discharged from Hospital | 4
Not completed — Death | 2
Not completed — Care Transferred to Another Physician | 2
Not completed — Discontinued and Changed to Iodoflex | 1
Not completed — Physician Decision | 2
Not completed — Surrounding Wound Erythematous | 1
Not completed — Machine Losing Vaccum | 1
Not completed — Patient Lived Too Far Away | 1
Not completed — Above Knee Amputation | 1
Not completed — Reason Not Reported By Site | 1

BASELINE CHARACTERISTICS:
Population: The decision to report the 2 studies with a single CSR was due to high levels of similarity in both the study designs and the products themselves; the individual study designs were largely similar with the same patient population criteria, study endpoints, and data capture requirements; and the products were identical in terms of their indications for use and therapeutic delivery of NPWT.
Groups:
- NPWT (Non-Grafted Sites): Application of NPWT therapy to the wound - subjects with a non-grafted wound site
  EZCARE/V1STA Negative Pressure Wound Therapy System: Vacuum Source and dressing kit that generates negative pressure over the wound.
- NPWT (Grafted Sites): Application of NPWT therapy to the wound - subjects with a grafted wound site
  EZCARE/V1STA Negative Pressure Wound Therapy System: Vacuum Source and dressing kit that generates negative pressure over the wound.
- Total: Total of all reporting groups
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites) | Total
Number analyzed (Participants) | 131 | 21 | 152
Age, Continuous [Mean (Standard Deviation); unit: years of age] — Population: Not all sites reported demographics information for all enrolled subjects.
  years of age
    number analyzed (Participants) | 126 | 21 | 147
    (all) | 60.5 (16.8) | 43.2 (16.2) | 58.0 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all sites reported demographics information for all enrolled subjects.
  Participants
    number analyzed (Participants) | 130 | 21 | 151
    Female | 61 | 5 | 66
    Male | 69 | 16 | 85
Treatment Setting [Count of Participants; unit: Participants]
  Long-term care/nursing home | 3 | 0 | 3
  Home | 29 | 2 | 31
  Hospital | 76 | 19 | 95
  Wound Clinic | 23 | 0 | 23
Patient Mobility [Count of Participants; unit: Participants]
  Walks Unaided | 50 | 12 | 62
  Walks with Aid | 30 | 5 | 35
  Walks Unaided/Walks with Aid | 0 | 1 | 1
  Chair Bound | 16 | 2 | 18
  Walks with Aid/Chair Bound | 1 | 0 | 1
  Bed Bound | 31 | 1 | 32
  Chair Bound/Bed Bound | 3 | 0 | 3
Medical History [Count of Participants; unit: Participants]
  Anemia: Current condition | 8 | 0 | 8
  Anemia: Prior condition | 3 | 0 | 3
  Anemia: Had condition, current/prior not given | 4 | 1 | 5
  Anemia: Never had the condition | 116 | 20 | 136
  Diabetes: Current condition | 26 | 4 | 30
  Diabetes: Prior condition | 2 | 0 | 2
  Diabetes: Had condition, current/prior not given | 23 | 1 | 24
  Diabetes: Never had the condition | 80 | 16 | 96
  Stroke/cardiovascular accident (CVA): Current condition | 3 | 0 | 3
  Stroke/cardiovascular accident (CVA): Prior condition | 7 | 0 | 7
  Stroke/cardiovascular accident (CVA): Had condition, current/prior not given | 7 | 0 | 7
  Stroke/cardiovascular accident (CVA): Never had the condition | 114 | 21 | 135
  Hypertension: Current condition | 29 | 2 | 31
  Hypertension: Prior condition | 2 | 0 | 2
  Hypertension: Had condition, current/prior not given | 27 | 1 | 28
  Hypertension: Never had the condition | 73 | 18 | 91
  Peripheral vascular disease: Current condition | 11 | 0 | 11
  Peripheral vascular disease: Prior condition | 1 | 0 | 1
  Peripheral vascular disease: Had condition, current/prior not given | 17 | 1 | 18
  Peripheral vascular disease: Never had the condition | 102 | 20 | 122
  Congestive heart failure: Current condition | 4 | 0 | 4
  Congestive heart failure: Prior condition | 2 | 1 | 3
  Congestive heart failure: Had condition, current/prior not given | 6 | 0 | 6
  Congestive heart failure: Never had the condition | 119 | 20 | 139
  Rheumatoid arthritis: Current condition | 2 | 0 | 2
  Rheumatoid arthritis: Prior condition | 0 | 0 | 0
  Rheumatoid arthritis: Had condition, current/prior not given | 5 | 0 | 5
  Rheumatoid arthritis: Never had the condition | 124 | 21 | 145
  Osteoarthritis: Current condition | 3 | 0 | 3
  Osteoarthritis: Prior condition | 0 | 0 | 0
  Osteoarthritis: Had condition, current/prior not given | 16 | 0 | 16
  Osteoarthritis: Never had the condition | 112 | 21 | 133
  Deep vein thrombosis (DVT): Current condition | 1 | 0 | 1
  Deep vein thrombosis (DVT): Prior condition | 1 | 0 | 1
  Deep vein thrombosis (DVT): Had condition, current/prior not given | 0 | 0 | 0
  Deep vein thrombosis (DVT): Never had the condition | 129 | 21 | 150
  Varicose veins: Current condition | 2 | 0 | 2
  Varicose veins: Prior condition | 1 | 0 | 1
  Varicose veins: Had condition, current/prior not given | 2 | 1 | 3
  Varicose veins: Never had the condition | 126 | 20 | 146
Wound Type [Count of Participants; unit: Participants]
  Surgical wound | 63 | 0 | 63
  Traumatic wound | 12 | 0 | 12
  Pressure ulcer | 34 | 0 | 34
  Diabetic foot ulcer | 15 | 0 | 15
  Leg ulcer | 4 | 0 | 4
  Graft site | 0 | 21 | 21
  Other wound | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Wounds Stratified by Wound Area for the Performance of EZCare/V1STA in Terms of Wound Progress Towards Closure in Wounds Deemed Suitable for Treatment With Negative Pressure Wound Therapy (NPWT) - Wound Area (Baseline Measurements)
Description: Evaluation was conducted to determine the extent of wound progression by the use of the NPWT EZCare/V1STA devices. Analysis of the amount of granulation tissue formation, successful management of exudate, and wound progression by reduction in area, volume, and depth were measured to assess improvement in wound healing. The wound was measured to assess wound area at Baseline.
Time Frame: Baseline
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects present at Baseline as provided by the site.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Groups:
- NPWT (Non-Grafted Sites); NPWT (Grafted Sites): Application of NPWT therapy to the wound
  EZCare/V1STA Negative Pressure Wound Therapy System: Vacuum Source and dressing kit that generates negative pressure over the wound.
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 127 | 21
Number analyzed (Wounds) | 127 | 21
Wounds
  <10 cm^2 wound area | 36 | 2
  10 cm^2 to <20 cm^2 wound area | 28 | 1
  >= 20 cm^2 wound area | 63 | 18

2. Primary Outcome: Number of Wounds Stratified by Change in Wound Area for the Performance of EZCare/V1STA in Terms of Wound Progress Towards Closure in Wounds Deemed Suitable for Treatment With Negative Pressure Wound Therapy (NPWT) - Wound Area (Follow-up Visits)
Description: Evaluation was conducted to determine the extent of wound progression by the use of the NPWT EZCare/V1STA devices. Analysis of wound progression by reduction in area was measured to assess improvement in wound healing. The wound was measured for change in wound area from Baseline compared to study discontinuation/withdrawal (up to 30 days of treatment plus a 7-day follow-up visit after discontinuation of NPWT).
Time Frame: Baseline to Treatment Discontinuation (up to 30 days of treatment plus an additional 7-day follow-up visit after treatment discontinuation)
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects showing measurable reduction in wound area from Baseline measurements at the specified time point visits.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 125 | 21
Number analyzed (Wounds) | 125 | 21
Wounds
  Wound Progression at Treatment Discontinuation by Baseline Wound Area <10 cm^2: number analyzed (Participants) | 36 | 2
  Wound Progression at Treatment Discontinuation by Baseline Wound Area <10 cm^2: number analyzed (Wounds) | 36 | 2
  Wound Progression at Treatment Discontinuation by Baseline Wound Area <10 cm^2: Healed/Closed | 5 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Area <10 cm^2: Progressing to closure/healing | 27 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Area <10 cm^2: Not progressing to closure/healing | 4 | 0
  Wound Progression at Treatment Discontinuation by Baseline Wound Area 10 cm^2 to <20 cm^2: number analyzed (Participants) | 27 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Area 10 cm^2 to <20 cm^2: number analyzed (Wounds) | 27 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Area 10 cm^2 to <20 cm^2: Healed/Closed | 7 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Area 10 cm^2 to <20 cm^2: Progressing to closure/healing | 18 | 0
  Wound Progression at Treatment Discontinuation by Baseline Wound Area 10 cm^2 to <20 cm^2: Not progressing to closure/healing | 2 | 0
  Wound Progression at Treatment Discontinuation by Baseline Wound Area >= 20 cm^2: number analyzed (Participants) | 62 | 18
  Wound Progression at Treatment Discontinuation by Baseline Wound Area >= 20 cm^2: number analyzed (Wounds) | 62 | 18
  Wound Progression at Treatment Discontinuation by Baseline Wound Area >= 20 cm^2: Healed/Closed | 4 | 4
  Wound Progression at Treatment Discontinuation by Baseline Wound Area >= 20 cm^2: Progressing to closure/healing | 51 | 13
  Wound Progression at Treatment Discontinuation by Baseline Wound Area >= 20 cm^2: Not progressing to closure/healing | 7 | 1

3. Primary Outcome: Number of Wounds Stratified by Wound Volume for the Performance of EZCare/V1STA in Terms of Wound Progress Towards Closure in Wounds Deemed Suitable for Treatment With NPWT - Wound Volume (Baseline Measurements)
Description: Evaluation was conducted to determine the extent of wound progression by the use of the NPWT EZCare/V1STA devices. Analysis of the amount of granulation tissue formation, successful management of exudate, and wound progression by reduction in area, volume, and depth were measured to assess improvement in wound healing. The wound was measured for wound volume at Baseline.
Time Frame: Baseline
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects present at Baseline.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 123 | 20
Number analyzed (Wounds) | 123 | 20
Wounds
  <20 cm^3 wound volume | 42 | 11
  20 cm^3 to <100 cm^3 wound volume | 51 | 5
  >= 100 cm^3 wound volume | 30 | 4

4. Primary Outcome: Number of Wounds Stratified by Change in Wound Volume for the Performance of EZCare/V1STA in Terms of Wound Progress Towards Closure in Wounds Deemed Suitable for Treatment With NPWT - Wound Volume (Follow-up Visits)
Description: Evaluation was conducted to determine the extent of wound progression by the use of the NPWT EZCare/V1STA devices. Analysis of the amount of wound progression by reduction in volume was measured to assess improvement in wound healing. The wound was measured for change in wound volume from Baseline compared to study treatment discontinuation/withdrawal (up to 30 days of treatment plus a 7-day follow-up visit after discontinuation of NPWT).
Time Frame: as for outcome 2
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects showing measurable reduction in wound volume from Baseline measurements at the specified time point visits.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 123 | 20
Number analyzed (Wounds) | 123 | 20
Wounds
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume <20 cm^3: number analyzed (Participants) | 42 | 11
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume <20 cm^3: number analyzed (Wounds) | 42 | 11
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume <20 cm^3: Healed/closed | 9 | 3
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume <20 cm^3: Progressing to closure/healing | 27 | 8
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume <20 cm^3: Not progressing to closure/healing | 6 | 0
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume 20 cm^3 to <100 cm^3: number analyzed (Participants) | 51 | 5
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume 20 cm^3 to <100 cm^3: number analyzed (Wounds) | 51 | 5
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume 20 cm^3 to <100 cm^3: Healed/closed | 5 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume 20 cm^3 to <100 cm^3: Progressing to closure/healing | 41 | 3
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume 20 cm^3 to <100 cm^3: Not progressing to closure/healing | 5 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume >= 100 cm^3: number analyzed (Participants) | 30 | 4
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume >= 100 cm^3: number analyzed (Wounds) | 30 | 4
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume >= 100 cm^3: Healed/closed | 2 | 1
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume >= 100 cm^3: Progressing to closure/healing | 26 | 3
  Wound Progression at Treatment Discontinuation by Baseline Wound Volume >= 100 cm^3: Not progressing to closure/healing | 2 | 0

5. Primary Outcome: Number of Wounds Stratified by Wound Depth for the Performance of EZCare/V1STA in Terms of Wound Progress Towards Closure in Wounds Deemed Suitable for Treatment With NPWT - Wound Depth (Baseline Measurements)
Description: Evaluation was conducted to determine the extent of wound progression by the use of the NPWT EZCare/V1STA devices. Analysis of wound progression by reduction in depth was measured to assess improvement in wound healing. The wound was measured for wound depth at Baseline.
Time Frame: Baseline
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects at Baseline.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 126 | 20
Number analyzed (Wounds) | 126 | 20
Wounds
  0 cm wound depth | 4 | 4
  >0 cm to <4 cm wound depth | 99 | 16
  4 cm to <8 cm wound depth | 19 | 0
  >= 8 cm wound depth | 4 | 0

6. Secondary Outcome: Number of Participants Stratified by General Performance Characteristics Assessed for EZCare/V1STA NPWT - Ease of Application and Removal Participant Questionnaire
Description: Clinician evaluations of the general performance characteristics included ease of application and removal, duration of wear time, and time for each dressing change were assessed. The ease of application and removal of the dressing were assessed at study treatment discontinuation (removal)/study withdrawal.
Time Frame: Up to 30 days of treatment plus an additional 7-day follow-up visit after treatment discontinuation
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represents the clinician assessments for all enrolled subjects at the time of satisfaction survey.
Measure: Count of Participants; unit: Participants
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 123 | 20
Participants
  Ease of Application of Dressing: Exceeds expectations | 64 | 6
  Ease of Application of Dressing: Satisfied | 56 | 13
  Ease of Application of Dressing: Dissatisfied | 3 | 1
  Ease of Removal of Dressing: Exceeds expectations | 65 | 6
  Ease of Removal of Dressing: Satisfied | 58 | 14
  Ease of Removal of Dressing: Dissatisfied | 0 | 0

7. Secondary Outcome: Number of Wounds Stratified by General Performance Characteristics Assessed for EZCare/V1STA NPWT - Duration of Wear Time
Description: Evaluation of the general performance characteristics included ease of application and removal, duration of wear time, and time for each dressing change were assessed. Duration of wear time was assessed based on the Baseline level of exudate.
Time Frame: Baseline up to 30 days of treatment plus an additional 7-day follow-up visit after treatment discontinuation
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects necessitating dressing changes based on level of exudate from wound at each time point.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 129 | 16
Number analyzed (Wounds) | 129 | 16
days
  Baseline Level of Exudate - None (duration of wear time): number analyzed (Participants) | 11 | 3
  Baseline Level of Exudate - None (duration of wear time): number analyzed (Wounds) | 11 | 3
  Baseline Level of Exudate - None (duration of wear time) | 2.8 (0.5) | 2.3 (2.1)
  Baseline Level of Exudate - Mild (duration of wear time): number analyzed (Participants) | 42 | 9
  Baseline Level of Exudate - Mild (duration of wear time): number analyzed (Wounds) | 42 | 9
  Baseline Level of Exudate - Mild (duration of wear time) | 2.9 (0.5) | 3.1 (1.2)
  Baseline Level of Exudate - Moderate (duration of wear time): number analyzed (Participants) | 57 | 4
  Baseline Level of Exudate - Moderate (duration of wear time): number analyzed (Wounds) | 57 | 4
  Baseline Level of Exudate - Moderate (duration of wear time) | 2.7 (0.5) | 2.6 (0.9)
  Baseline Level of Exudate - Heavy (duration of wear time): number analyzed (Participants) | 19 | 0
  Baseline Level of Exudate - Heavy (duration of wear time): number analyzed (Wounds) | 19 | 0
  Baseline Level of Exudate - Heavy (duration of wear time) | 2.7 (0.7) |
  Overall Duration of Wear Time by Level of Exudate | 2.8 (0.5) | 2.8 (1.3)

8. Secondary Outcome: Number of Dressing Changes Stratified by General Performance Characteristics Assessed for EZCare/V1STA NPWT - Time for Each Dressing Change
Description: Evaluation of the general performance characteristics included ease of application and removal, duration of wear time, and time for each dressing change were assessed. Based on the number of dressing changes performed throughout the study on all enrolled subjects, the average time it took to change each dressing was analyzed.
Time Frame: Baseline up to 30 days of treatment plus an additional 7-day follow-up visit after treatment discontinuation
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent how many minutes on average it took to change the dressing.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Number of Dressing Changes
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 131 | 21
Number analyzed (Number of Dressing Changes) | 827 | 36
minutes | 19.7 (10.4) | 14.2 (8.4)

9. Secondary Outcome: Number of Wounds Stratified by Pain Level for the Analysis of Wound Pain Over the Treatment Period
Description: Evaluation of wound pain was determined by assessing pain over the treatment period (unrelated to dressing application or removal).
Time Frame: Baseline up to 30 days of treatment plus an additional 7-day follow-up visit after treatment discontinuation
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects' survey responses at each time point.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 130 | 21
Number analyzed (Wounds) | 813 | 37
Wounds
  Level of Pain in the Past Week at Baseline: number analyzed (Wounds) | 130 | 21
  Level of Pain in the Past Week at Baseline: None | 58 | 4
  Level of Pain in the Past Week at Baseline: Mild | 42 | 11
  Level of Pain in the Past Week at Baseline: Moderate | 24 | 5
  Level of Pain in the Past Week at Baseline: Severe | 6 | 1
  Level of Pain in the Past Week at Treatment Discontinuation: number analyzed (Wounds) | 130 | 21
  Level of Pain in the Past Week at Treatment Discontinuation: None | 101 | 12
  Level of Pain in the Past Week at Treatment Discontinuation: Mild | 23 | 8
  Level of Pain in the Past Week at Treatment Discontinuation: Moderate | 6 | 1
  Level of Pain in the Past Week at Treatment Discontinuation: Severe | 0 | 0
  Level of Pain in the Past Week at 7-Day Post Treatment Follow-up Visit: number analyzed (Participants) | 73 | 17
  Level of Pain in the Past Week at 7-Day Post Treatment Follow-up Visit: number analyzed (Wounds) | 73 | 17
  Level of Pain in the Past Week at 7-Day Post Treatment Follow-up Visit: None | 63 | 11
  Level of Pain in the Past Week at 7-Day Post Treatment Follow-up Visit: Mild | 7 | 5
  Level of Pain in the Past Week at 7-Day Post Treatment Follow-up Visit: Moderate | 3 | 1
  Level of Pain in the Past Week at 7-Day Post Treatment Follow-up Visit: Severe | 0 | 0
  Level of Pain at Dressing Removal Overall: None | 666 | 18
  Level of Pain at Dressing Removal Overall: Mild | 108 | 17
  Level of Pain at Dressing Removal Overall: Moderate | 37 | 1
  Level of Pain at Dressing Removal Overall: Severe | 2 | 1

10. Secondary Outcome: Number of Wounds Stratified by Level of Odor for Analysis Over the Treatment Period
Description: Evaluation of wound odor was assessed over the duration of the treatment period at each respective time point.
Time Frame: Baseline up to 30 days of treatment plus an additional 7-day follow-up visit after treatment discontinuation
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects participating in the survey at each specified time point.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 131 | 21
Number analyzed (Wounds) | 131 | 21
Wounds
  Level of Wound Odor at Baseline: None | 80 | 18
  Level of Wound Odor at Baseline: Slight | 35 | 3
  Level of Wound Odor at Baseline: Moderate | 10 | 0
  Level of Wound Odor at Baseline: Strong | 6 | 0
  Level of Wound Odor at Treatment Discontinuation: number analyzed (Participants) | 130 | 20
  Level of Wound Odor at Treatment Discontinuation: number analyzed (Wounds) | 130 | 20
  Level of Wound Odor at Treatment Discontinuation: None | 107 | 19
  Level of Wound Odor at Treatment Discontinuation: Slight | 19 | 1
  Level of Wound Odor at Treatment Discontinuation: Moderate | 2 | 0
  Level of Wound Odor at Treatment Discontinuation: Strong | 2 | 0
  Level of Wound Odor at 7-Day Post Treatment Follow-up Visit: number analyzed (Participants) | 66 | 16
  Level of Wound Odor at 7-Day Post Treatment Follow-up Visit: number analyzed (Wounds) | 66 | 16
  Level of Wound Odor at 7-Day Post Treatment Follow-up Visit: None | 59 | 15
  Level of Wound Odor at 7-Day Post Treatment Follow-up Visit: Slight | 5 | 1
  Level of Wound Odor at 7-Day Post Treatment Follow-up Visit: Moderate | 2 | 0
  Level of Wound Odor at 7-Day Post Treatment Follow-up Visit: Strong | 0 | 0

11. Primary Outcome: Number of Wounds Stratified by Improvement in Wound Depth for the Performance of EZCare/V1STA in Terms of Wound Progress Towards Closure in Wounds Deemed Suitable for Treatment With NPWT - Wound Depth (Follow-up Visits)
Description: Evaluation was conducted to determine the extent of wound progression by the use of the NPWT EZCare/V1STA devices. Analysis of wound progression by improvement in depth was measured to assess improvement in wound healing. The wound was measured for change in depth from Baseline to study treatment discontinuation/withdrawal.
Time Frame: Baseline up to 20 weeks post initial treatment
Population: The study was further divided into subgroups of subjects with a grafted wound site or subjects with a non-grafted wound site to compare wound types. The data presented represent the enrolled subjects showing measurable improvement in wound depth from Baseline measurements at the specified time point visits.
Measure: Mean (Standard Deviation); unit: percentage of improvement in depth
Units Other Than Participants: Wounds
Arm/Group | NPWT (Non-Grafted Sites) | NPWT (Grafted Sites)
Number analyzed (Participants) | 112 | 15
Number analyzed (Wounds) | 112 | 15
percentage of improvement in depth
  Wound Duration <1 Week: number analyzed (Participants) | 3 | 2
  Wound Duration <1 Week: number analyzed (Wounds) | 3 | 2
  Wound Duration <1 Week | 42.2 (23.4) | 70 (42.4)
  Wound Duration 1 - <4 Weeks: number analyzed (Participants) | 34 | 5
  Wound Duration 1 - <4 Weeks: number analyzed (Wounds) | 34 | 5
  Wound Duration 1 - <4 Weeks | 47.8 (68.1) | 38.8 (46.9)
  Wound Duration 4 - <20 Weeks: number analyzed (Participants) | 45 | 6
  Wound Duration 4 - <20 Weeks: number analyzed (Wounds) | 45 | 6
  Wound Duration 4 - <20 Weeks | 48.8 (33.9) | 29.1 (15.4)
  Wound Duration >=20 Weeks: number analyzed (Participants) | 30 | 2
  Wound Duration >=20 Weeks: number analyzed (Wounds) | 30 | 2
  Wound Duration >=20 Weeks | 41.0 (49.7) | 29.1 (15.4)

ADVERSE EVENTS:
Time Frame: Baseline through end of study treatment (30 days of treatment plus 7-day follow-up assessment).
Description: While starting out as two individual studies (EZCare CIME 012 and V1STA CIME 010), these studies were combined and analyzed together as one set of results due to high levels of similarity in both the study designs and the products themselves.
Arm/Group | Negative Pressure Wound Therapy
All-Cause Mortality (participants affected / at risk) | 2/153
Serious Adverse Events (participants affected / at risk) | 2/153
Other Adverse Events (participants affected / at risk) | 1/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Pressure Wound Therapy (N=153)
Natural Causes (General disorders) | 1 (1) — Investigator stated death was expected due to age and comorbidities, not related to the product.
Alcoholic Liver Disease (Hepatobiliary disorders) | 1 (1) — Investigator reported multiorgan failure due to alcoholic liver disease, not related to the product.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Pressure Wound Therapy (N=153)
Peri-wound maceration and inflammation (Skin and subcutaneous tissue disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
While starting out as two individual studies (EZCare CIME 012 and V1STA CIME 010), these studies were combined and analyzed together as one set of results due to high levels of similarity in both the study designs and the products themselves. This was a non-controlled study delivering a global dataset with potential bias towards North America. V1STA was set up as a global study and EZCare was focused on the USA and Canada. This resulted in 108 of the 153 patients being from North America.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days